CLINICAL TRIAL: NCT02823015
Title: Acute Pain Trajectories as a Predictive Factor for Persistent Pain After Breast Cancer Surgery
Brief Title: Acute Pain Trajectories and Persistent Pain After Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ANES-AS-002
Record Dates: First submitted 2016-05-30; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study population: The study population consists of adult surgery patients, scheduled for breast cancer surgery at St-Luc University Hospital.

SUMMARY:
Persistent pain after breast cancer surgery (PPBCS) is a significant clinical problem, affecting between 25 and 50% of patients. Several factors are associated with the development of PPBCS, including acute postoperative pain. The analysis of pain trajectories through mixed model modeling is an alternative to static pain measures, improving precision and providing information on the time course of pain resolution. Our aim was to investigate if the characteristics of pain trajectories during the first postoperative week are correlated with the persistence of pain 3 months after breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for breast cancer surgery
* General anesthesia

Exclusion Criteria:

* Previous breast surgery
* Reconstructive surgery scheduled during follow-up
* Day-surgery patients
* Inability to understand the questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females, scheduled for breast cancer surgery
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Presence of pain 3 months after surgery, assessed with the Brief Pain Inventory questionnaire. Yes/No | 3 months

SECONDARY OUTCOMES:
Acute pain trajectories (7 days) after surgery | One postoperative week
  The pain trajectory is the vector of 7 verbal numerical pain scores (from 0 to 10) recorded in a pain diary over the first 7 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Steyaert, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Woluwé-St-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: Undecided